CLINICAL TRIAL: NCT01601938
Title: Effects of Selenium Replacement on Prognosis of Severe Sepsis and Septic Shock Patients and Their Initial Serum Selenium Level: a Randomized, Double-blind Placebo Controlled Phase 2 Study
Brief Title: Selenium Replacement and Serum Selenium Level in Severe Sepsis and Septic Shock Patients
Acronym: SEREAL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: We failed to obtain study drugs from the company
Sponsor: Gil Joon Suh (Other)
Collaborators: Biosyn (Industry); Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Gil Joon Suh, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUHEM-SEREAL-12-0001
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Sepsis; Shock, Septic
Keywords: Sepsis; Shock, Septic; Selenium; Survival
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selenium (Experimental): 500 mcg of selenium (10mL) daily for 7 days
  Interventions: Dietary Supplement: selenium replacement
- Placebo (Placebo Comparator): Placebo 10 mL (delivered from biosyn) for 7 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: selenium replacement — Selenium 500 mcg (10 mL) mixed to 230 mL of normal saline will be infused continuously per day (10 mL/hour). Study drugs will be infused for 7 days.
  Other Names: Selenase T pro injectione
  Arms: Selenium
Dietary Supplement: Placebo — placebo (10 mL) mixed to 230 mL of normal saline will be infused continuously per day (10 mL/hour). Study drugs will be infused for 7 days.
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
This study will be performed to determine whether selenium replacement reduces 28-day mortality of severe sepsis and septic shock patients, and to investigate whether selenium replacement contributes differently to the mortality reduction of the patients according to their initial serum selenium level.

DETAILED DESCRIPTION:
This study is a single center, randomized, double-blind, placebo controlled trial.

After the diagnosis of severe sepsis and septic shock, enrolled patients will be randomized. Then, selenium or placebo will be intravenously administered to them for 7 days. Hemodynamic and laboratory data will be recorded for 7 days and additional serum samples will be obtained at 0, 24, 72, and 168 hours post-treatment and stored. Mortality will be observed for 28 days.

An interim analysis will be conducted by the independent data safety monitoring board.

Serum selenium levels will be measured from the stored serum samples after the study completion.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* clinical diagnosis of severe sepsis or septic shock

Exclusion Criteria:

* pregnancy or breast feeding
* age younger than 18
* advanced directive state to withhold treatment
* known allergy to selenium
* CPR or death within 24 hours after the diagnosis of severe sepsis or septic shock
* advanced malignancy without further treatment plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  All cause mortality occurs within 28 days.

SECONDARY OUTCOMES:
ICU length of stay | 3 months
  After 3 months from enrollment, the participant's ICU length of stay will be evaluated.
Mortality at hospital discharge | 3 months
  After 3 months from enrollment, the participant's in hospital mortality will be evaluated.
Development of the new infection | 3 months
  After 3 months from enrollment, the development of new infection of the participant during the hospitalization will be evaluated.
Serum selenium level | At 0, 24, 72, 168 hours post-enrollment
  After study completion, serum selenium level will be measured from stored samples. Then, we will investigate whether selenium replacement contributes differently to the mortality reduction of the enrolled patients according to their initial serum selenium level.
Ventilator days | 3 months
  After 3 months from enrollment, total numbers of ventilator days of the participant during the hospitalization will be evaluated.
Renal replacement therapy days | 3 months
  After 3 months from enrollment, the days of renal replacement therapy of the participant during the hospitalization will be evaluated.
Oxidative stress marker | At 0, 24, 72, 168 hours post-enrollment
  After study completion, serum glutathione peroxidase, reduced glutathione, NADPH, and MDA will be measured from stored samples.
Changes in severity scores | 7 days
  APACHE II score, SOFA score, and SAPS II will be calculated at 1, 3, 7 days
3-month mortality | 3 months post-enrollment
Inflammatory markers | At 0, 24, 72, 268 hours post-enrollment
  After study completion, serum cytokines, CRP, and chemokines will be measured from stored samples.
Vasopressor days | 3 months
  Days of dopamine, norepinephrine, dobutamine, vasopressin, and epinephrine will be investigated

CONTACTS AND LOCATIONS:
Overall Officials: Gil Joon Suh, professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Angstwurm MW, Engelmann L, Zimmermann T, Lehmann C, Spes CH, Abel P, Strauss R, Meier-Hellmann A, Insel R, Radke J, Schuttler J, Gartner R. Selenium in Intensive Care (SIC): results of a prospective randomized, placebo-controlled, multiple-center study in patients with severe systemic inflammatory response syndrome, sepsis, and septic shock. Crit Care Med. 2007 Jan;35(1):118-26. doi: 10.1097/01.CCM.0000251124.83436.0E. PMID 17095947
- [Background] Andrews PJ, Avenell A, Noble DW, Campbell MK, Croal BL, Simpson WG, Vale LD, Battison CG, Jenkinson DJ, Cook JA; Scottish Intensive care Glutamine or seleNium Evaluative Trial Trials Group. Randomised trial of glutamine, selenium, or both, to supplement parenteral nutrition for critically ill patients. BMJ. 2011 Mar 17;342:d1542. doi: 10.1136/bmj.d1542. PMID 21415104
- [Background] Forceville X, Laviolle B, Annane D, Vitoux D, Bleichner G, Korach JM, Cantais E, Georges H, Soubirou JL, Combes A, Bellissant E. Effects of high doses of selenium, as sodium selenite, in septic shock: a placebo-controlled, randomized, double-blind, phase II study. Crit Care. 2007;11(4):R73. doi: 10.1186/cc5960. PMID 17617901